CLINICAL TRIAL: NCT00548938
Title: A Phase II Study of Gliadel, Concomitant Temozolomide and Radiation, Followed by Metronomic Therapy With Temozolomide for Newly Diagnosed Malignant High Grade Glioma
Brief Title: Gliadel Wafer, Temozolomide and Radiation Therapy for Newly Diagnosed GBM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator has left the institution
Sponsor: Methodist Healthcare (Other)
Responsible Party: Allen Sills, MD, Methodist Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHIRB #2007-040
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Glioblastoma Multiforme; High-Grade Glioma
Keywords: Brain Tumor; GBM; Glioblastoma Multiforme; Giladel; Temozolomide
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Carmustine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gliadel wafer — Implanted at surgery
Drug: Temozolomide — During External Beam Radiation
Radiation: External Beam Radiation Therapy — 60 Gy

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the combination of Gliadel wafers plus surgery and limited field radiation therapy with concomitant temozolomide followed by temozolomide given at an extended dose schedule (metronomic schedule) in patients undergoing initial surgery for newly-diagnosed high grade glioma.

DETAILED DESCRIPTION:
The patient population in this Phase II clinical trial will be patients with newly diagnosed high-grade glioma undergoing initial surgery. Patients will receive Surgery + Gliadel® wafer implantation + Limited Field Radiation Therapy with concomitant daily temozolomide (75 mg/m2) followed by monthly temozolomide given at the same dose (75 mg/m2 per day for 21 days each month.

Patients will have up to 8 wafers implanted into the tumor resection cavity (depending upon its size) after maximal tumor resection. Between Study Days 14 and 45 all patients will begin a standard course of post-operative limited field radiation therapy to the tumor site and a surrounding margin. Temozolomide will be administered concomitantly with radiation at a daily dose of 75 mg/m2 daily (7 days/week) and then beginning no later than 30 days following completion of radiation therapy on a 75 mg/m2 daily dose given 21 days out of each month for a total of up to 18 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, must be between ages 18-72
* Patients must have radiographic evidence on cranial magnetic resonance imaging (MRI) of a single, contrast-enhancing unilateral supratentorial cerebral tumor suggestive of high-grade glioma
* Surgical treatment within 4 weeks of the baseline MRI is indicated
* Karnofsky Performance Score of 60 or higher
* Patients must have a pathological diagnosis of high-grade (IV) malignant glioma
* Patients must be willing to use a barrier method of contraception if fertile or if of childbearing potential for up to 2 years after wafer implantation and be counseled regarding the unknown, and potentially harmful, risks to the embryo or fetus while treated on this study

Exclusion Criteria:

* Patients who have had prior cytoreductive surgery for high-grade glioma (patients who have had a diagnostic stereotactic biopsy are eligible)
* Patients with more than one focus of tumor or tumor crossing the midline as assessed by coronal cranial MRI scan
* Concomitant significant life-threatening disease from which the patient could reasonably be expected to die within the first 12 months of the study
* Known hypersensitivity reactions to temozolomide, nitrosoureas or any components of the Gliadel wafer
* Prior CNS radiotherapy
* Patients who have received any prior chemotherapy for malignant glioma prior to the baseline evaluation or patients who are currently being treated with chemotherapeutic agents
* Patients with fewer than 100,000 platelets per mm3 or fewer than 3,500 leukocytes per mm3
* Liver function tests greater than or equal to 2.5 times the upper limit of normal (transaminases (SGOT, SGPT), total bilirubin, alkaline phosphatase)
* Serum creatinine equal to or greater than 1.5 times the upper limit of normal, blood urea nitrogen (BUN) equal to or greater than 2.5 times the upper limit of normal
* Pregnancy, or lactating females or females of childbearing potential not employing adequate contraception
* Participation in any other investigational protocol in the prior twelve months for any type of malignancy
* Psychological, familial, sociological or geographical conditions which do not permit adequate medical follow-up and compliance with the study protocol

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of Gliadel wafer + radiation + temozolomide in patients with newly diagnosed high grade glioma undergoing surgery as determined by time to disease progression. | 2 years

SECONDARY OUTCOMES:
Median, one year and overall survival rate. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Allen K Sills, MD, Principal Investigator — Methodist University Hospital
Locations (1):
- Methodist University Hospital, Memphis, Tennessee, United States